CLINICAL TRIAL: NCT02412306
Title: A Phase 1b/2 Study of Blinatumomab in Japanese Subjects With Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia (ALL) (Horai Study)
Brief Title: Study of Blinatumomab in Japanese Patients With Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Amgen Astellas Biopharma K.K. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20130265
Record Dates: First submitted 2015-03-12; First posted 2015-04-09 (Estimated); Results first posted 2020-01-10 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Relapsed Refractory B Precursor Acute Lymphoblastic Leukemia
Keywords: Amgen
MeSH Terms: interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Blinatumomab 9-28 µg/day Phase 1b Adult Population (Experimental): Participants received blinatumomab by continuous intravenous (CIV) infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose for adults was 9 µg/day for the first week of cycle 1, escalated to 28 µg/day starting from Week 2 and all cycles thereafter.
  Interventions: Drug: Blinatumomab
- Blinatumomab 5-15 µg/m^2/day Phase 1b Pediatric Population (Experimental): Participants received blinatumomab by CIV infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. For pediatric participants the initial dose was 5 µg/m²/day for the first week of cycle 1, escalated to 15 µg/m²/day starting from week 2 and all cycles thereafter.
  Interventions: Drug: Blinatumomab
- Blinatumomab 9-28 µg/day Phase 2 Adult Population (Experimental): Participants received blinatumomab by CIV infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose for adults was 9 µg/day for the first week of cycle 1, escalated to 28 µg/day starting from Week 2 and all cycles thereafter.
  Interventions: Drug: Blinatumomab
- Blinatumomab 9-28 µg/day Adult Expansion Population (Experimental): Participants received blinatumomab by CIV infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose for adults was 9 µg/day for the first week of cycle 1, escalated to 28 µg/day starting from Week 2 and all cycles thereafter.
  Interventions: Drug: Blinatumomab
- Blinatumomab 5-15 µg/m^2/day Pediatric Expansion Population (Experimental): Participants received blinatumomab by CIV infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. For pediatric participants the initial dose was 5 µg/m²/day for the first week of cycle 1, escalated to 15 µg/m²/day starting from week 2 and all cycles thereafter.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Continuous intravenous infusion over four weeks per treatment cycle
  Other Names: Blincyto®

SUMMARY:
This is an open-label, combined 2-part multicenter study to evaluate the efficacy, safety, and tolerability of blinatumomab in adult and pediatric Japanese patients with relapsed/refractory B-precursor ALL.

DETAILED DESCRIPTION:
The Phase 1b part will investigate the safety, efficacy, pharmacokinetics (PK) and pharmacodynamics (PD) of blinatumomab to determine the maximum tolerated dose (MTD) in both adult and pediatric Japanese patients with relapsed/refractory B-precursor ALL. The Phase 2 part will assess the safety and efficacy of the recommended dose level of blinatumomab identified in the Phase 1b portion of the study in the adult study population.

In June 2017 protocol amendment 4 extended the study to include an expansion cohort of approximately 65 participants to investigate the safety of blinatumomab in participants who did not participate in Phase 1b or Phase 2 of the study. Adult and pediatric patients in the expansion cohort may receive up to 5 cycles of investigational blinatomumab and may receive commercial blinatomumab after a minimum of 2 cycles of the investigational drug.

ELIGIBILITY:
Adult Subjects Key Inclusion Criteria:

* Age ≥ 18 years old at enrollment
* Subjects with Philadelphia-negative B-precursor ALL, with any of the following:

  * Relapsed or refractory after first line therapy with first remission duration ≤ 12 months; or
  * Relapsed or refractory after first salvage therapy; or
  * Relapsed or refractory within 12 months of allogeneic hematopoietic stem cell transplant (alloHSCT)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
* Greater than 5% blasts in bone marrow

Pediatric Subjects Key Inclusion Criteria:

* Age < 18 years old at enrollment
* Relapsed/refractory disease, defined as one of the following:

  * second or later bone marrow relapse;
  * any marrow relapse after alloHSCT; or
  * Refractory to other treatments:

    * For subjects in first relapse: failure to achieve a complete response (CR) following a full standard reinduction chemotherapy regimen
    * For subjects who have not achieved a first remission: failure to achieve remission following a full standard induction regimen
* Greater than 5% blasts in bone marrow
* Karnofsky performance status ≥ 50% for subjects ≥ 16 years
* Lansky performance status ≥ 50% for subjects < 16 years

Key Exclusion Criteria

* Subjects with Burkitt´s Leukemia according to World Health Organization (WHO) classification
* History or presence of clinically relevant central nervous system (CNS) pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis; with the exception of well-controlled CNS leukemia
* Active ALL in the CNS or testes
* Current autoimmune disease or history of autoimmune disease with potential CNS involvement
* Autologous HSCT within 6 weeks prior to start of blinatumomab treatment
* AlloHSCT within 12 weeks prior to start of blinatumomab treatment
* Any active acute Graft-versus-Host Disease (GvHD) grade 2-4 according to Glucksberg criteria or active chronic GvHD requiring systemic treatment

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (16):
- Japan (16):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Gunmaken Saiseikai Maebashi Hospital, Maebashi, Gunma
  - Sapporo Hokuyu Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Kanagawa Childrens Medical Center, Yokohama, Kanagawa
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Okayama University Hospital, Okayama, Okayama-ken
  - Osaka City General Hospital, Osaka, Osaka
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - Saitama Childrens Medical Center, Saitama-shi, Saitama
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - National Center for Child Health and Development, Setagaya-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Horibe K, Morris JD, Tuglus CA, Dos Santos C, Kalabus J, Anderson A, Goto H, Ogawa C. A phase 1b study of blinatumomab in Japanese children with relapsed/refractory B-cell precursor acute lymphoblastic leukemia. Int J Hematol. 2020 Aug;112(2):223-233. doi: 10.1007/s12185-020-02907-9. Epub 2020 Jun 20. PMID 32564243
- [Background] Kiyoi H, Morris JD, Oh I, Maeda Y, Minami H, Miyamoto T, Sakura T, Iida H, Tuglus CA, Chen Y, Dos Santos C, Kalabus J, Anderson A, Hata T, Nakashima Y, Kobayashi Y. Phase 1b/2 study of blinatumomab in Japanese adults with relapsed/refractory acute lymphoblastic leukemia. Cancer Sci. 2020 Apr;111(4):1314-1323. doi: 10.1111/cas.14322. Epub 2020 Feb 11. PMID 31971321
- [Background] Kobayashi Y, Oh I, Miyamoto T, Lee WS, Iida H, Minami H, Maeda Y, Jang JH, Yoon SS, Yeh SP, Tran Q, Morris J, Franklin J, Kiyoi H. Efficacy and safety of blinatumomab: Post hoc pooled analysis in Asian adults with relapsed/refractory B-cell precursor acute lymphoblastic leukemia. Asia Pac J Clin Oncol. 2022 Jun;18(3):311-318. doi: 10.1111/ajco.13609. Epub 2021 Jun 29. PMID 34185953
- [Background] Goto H, Ogawa C, Iida H, Horibe K, Oh I, Takada S, Maeda Y, Minami H, Nakashima Y, Morris JD, Kormany W, Chen Y, Miyamoto T. Safety and Efficacy of Blinatumomab in Japanese Adult and Pediatric Patients with Relapsed/Refractory B-Cell Precursor Acute Lymphoblastic Leukemia: Final Results from an Expansion Cohort. Acta Haematol. 2022;145(6):592-602. doi: 10.1159/000525835. Epub 2022 Jul 5. PMID 35790143
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 16 centers in Japan. Cohort enrollment periods were: adult phase 1b, from 04 Jun 2015 to 13 Jan 2016; pediatric phase 1b, from 17 Feb 2016 to 20 Jun 2016; adult phase 2, from 11 Apr 2016 to 12 Jun 2017; adult expansion cohort, from 04 Dec 2017 to 13 Nov 2018; pediatric expansion cohort, from 05 Nov 2017 to 05 Sep 2018.
Pre-assignment Details: After a 2-week screening and pre-phase period, participants were treated in an open-label phase 1b part (adult or pediatric), a phase 2 part (adult), or in an expansion cohort (adult or pediatric).
Groups:
- Phase 1b: Blinatumomab 9/28 μg/Day (Adults): Participants received blinatumomab by continuous intravenous (CIV) infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose was 9 μg/day for the first week of cycle 1, escalated to 28 μg/day starting from week 2 and all cycles thereafter.
- Phase 1b: Blinatumomab 5/15 µg/m²/Day (Pediatric): Participants received blinatumomab by CIV over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose was 5 µg/m²/day for the first week of cycle 1, escalated to 15 µg/m²/day starting from week 2 and all cycles thereafter.
- Phase 2: Blinatumomab 9/28 μg/Day (Adults); Expansion Cohort: Blinatumomab 9/28 μg/Day (Adults): Participants received blinatumomab by continuous intravenous infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose was 9 μg/day for the first week of cycle 1, escalated to 28 μg/day starting from Week 2 and all cycles thereafter.
- Expansion Cohort: Blinatumomab 5/15 µg/m²/Day (Pediatric): Participants received blinatumomab by continuous intravenous infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose was 5 µg/m²/day for the first week of cycle 1, escalated to 15 µg/m²/day starting from week 2 and all cycles thereafter.
Period: Overall Study
Arm/Group | Phase 1b: Blinatumomab 9/28 μg/Day (Adults) | Phase 1b: Blinatumomab 5/15 µg/m²/Day (Pediatric) | Phase 2: Blinatumomab 9/28 μg/Day (Adults) | Expansion Cohort: Blinatumomab 9/28 μg/Day (Adults) | Expansion Cohort: Blinatumomab 5/15 µg/m²/Day (Pediatric)
Started | 5 | 9 | 21 | 14 | 17
Completed | 0 | 1 | 5 | 14 | 15
Not Completed | 5 | 8 | 16 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Death | 5 | 7 | 15 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Phase 1b: Blinatumomab 9/28 μg/Day (Adults): Participants received blinatumomab by CIV infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose was 9 μg/day for the first week of cycle 1, escalated to 28 μg/day starting from week 2 and all cycles thereafter.
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Blinatumomab 9/28 μg/Day (Adults) | Phase 1b: Blinatumomab 5/15 µg/m²/Day (Pediatric) | Phase 2: Blinatumomab 9/28 μg/Day (Adults) | Expansion Cohort: Blinatumomab 9/28 μg/Day (Adults) | Expansion Cohort: Blinatumomab 5/15 µg/m²/Day (Pediatric) | Total
Number analyzed (Participants) | 5 | 9 | 21 | 14 | 17 | 66
Age, Customized [Count of Participants; unit: Participants]
  < 2 years | 0 | 0 | 0 | 0 | 1 | 1
  2 to 6 years | 0 | 0 | 0 | 0 | 5 | 5
  7 to 17 years | 0 | 9 | 0 | 0 | 11 | 20
  18 to 34 years | 1 | 0 | 6 | 5 | 0 | 12
  35 to 54 years | 1 | 0 | 14 | 6 | 0 | 21
  55 to 64 years | 2 | 0 | 1 | 1 | 0 | 4
  ≥ 65 years | 1 | 0 | 0 | 2 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 12 | 9 | 8 | 38
  Male | 1 | 4 | 9 | 5 | 9 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 5 | 9 | 21 | 14 | 17 | 66

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose-limiting Toxicities
Description: Dose-limiting toxicities (DLTs) were defined as any Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 grade ≥ 3 adverse event related to blinatumomab, excluding specific CTCAE grade ≥ 3 adverse events considered consistent with the current known safety profile of blinatumomab, CTCAE grade ≥ 3 fever or infection, and laboratory parameters of CTCAE grade ≥ 3 not considered clinically relevant and/or responding to routine medical management.
Time Frame: Days 1 to 14
Population: Phase 1b participants in who received any infusion of blinatumomab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Blinatumomab 9/28 μg/Day (Adults) | Phase 1b: Blinatumomab 5/15 µg/m²/Day (Pediatric)
Number analyzed (Participants) | 5 | 9
Participants | 0 | 0

2. Primary Outcome: Phase 2: Percentage of Participants With a Best Response of Complete Remission or Complete Remission With Only Partial Hematological Recovery Within 2 Cycles of Treatment
Description: Hematological assessments were performed from bone marrow biopsy samples. All hematological assessments of bone marrow were reviewed in a central reference laboratory.
  Hematological remissions were defined by the following criteria:
  * Complete Remission (CR) is defined as ≤ 5% blasts in the bone marrow, no evidence of disease, and full recovery of peripheral blood counts: platelets > 100,000/µl and absolute neutrophil count (ANC) > 1,000/µl.
  * Complete Remission With Partial Hematological Recovery (CRh*) is defined as ≤ 5% blasts in the bone marrow, no evidence of disease, and partial recovery of peripheral blood counts: platelets > 50,000/µl and ANC > 500/µl.
Time Frame: Within the first 2 cycles of treatment, 12 weeks
Population: Phase 2 participants who received any infusion of blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Blinatumomab 9/28 μg/Day (Adults)
Number analyzed (Participants) | 21
percentage of participants | 38.1 [18.1 to 61.6]

3. Secondary Outcome: Phase 1b Adults: Percentage of Participants With a Best Response of Complete Remission or Complete Remission With Only Partial Hematological Recovery Within 2 Cycles of Treatment
Description: as for outcome 2
Time Frame: Within the first 2 cycles of treatment, 12 weeks
Population: Phase 1b adult participants who received any infusion of blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b: Blinatumomab 9/28 μg/Day (Adults)
Number analyzed (Participants) | 5
percentage of participants | 80.0 [28.4 to 99.5]

4. Secondary Outcome: Phase 1b Pediatric: Percentage of Participants With M1 Remission Within 2 Cycles of Treatment
Description: M1 remission for pediatric participants was defined as ≤ 5% blasts (M1 bone marrow) in the bone marrow and no evidence of disease.
Time Frame: The first 2 cycles of treatment, 12 weeks
Population: Phase 1b pediatric participants who received any infusion of blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b: Blinatumomab 5/15 µg/m²/Day (Pediatric)
Number analyzed (Participants) | 9
percentage of participants | 55.6 [21.2 to 86.3]

5. Secondary Outcome: Phase 1b and Phase 2: Duration of Response
Description: Duration of response was calculated from the date of bone marrow aspiration when response (CR/CRh*) was detected for the first time during the first 2 cycles of treatment until the earlier of the following events:
  * the date of bone marrow aspiration at which hematological relapse or progressive disease (PD) was first detected,
  * the date of diagnosis on which the hematological or extra medullary relapse was documented,
  * the date of death if patient died due to PD
  * the date of end of induction phase if primary reason for treatment termination was hematological or extramedullary relapse.
  For a responder who did not report an event and was alive during the study, the end date of duration (censoring) was based on the date of the last available bone marrow aspiration prior to the data cutoff date for the analysis. Participants with response who did not report an event and who died due to reasons other than PD, were censored on the date of death, with death treated as a competing risk.
Time Frame: Median (minimum [min], maximum [max]) follow-up time was 6.3 (2.4, 13.6) months for Phase 1b and 26.7 (3.0, 28.5) months for Phase 2.
Population: Phase 1b and Phase 2 participants who received any infusion of blinatumomab and achieved CR/CRh* during the first 2 cycles of treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b: Blinatumomab 9/28 μg/Day (Adults) | Phase 1b: Blinatumomab 5/15 µg/m²/Day (Pediatric) | Phase 2: Blinatumomab 9/28 μg/Day (Adults)
Number analyzed (Participants) | 4 | 5 | 8
months | 13.0 [4.2 to 19.7] | 2.3 [1.1 to 6.8] | 13.1 [3.5 to 20.7]

6. Secondary Outcome: Phase 1b and Phase 2: Relapse-free Survival
Description: Relapse-free survival (RFS) was defined for participants who achieved a response (CR/CRh*) during the first 2 cycles of treatment. RFS was calculated from the date of bone marrow aspiration when response was detected for the first time to the date of bone marrow aspiration at which hematological relapse was first detected or the date of diagnosis on which the hematological or extra medullary relapse was documented or the date of death due to any cause, whichever was earlier. Participants who did not experience hematological relapse and did not die were censored on the date of the last available bone marrow aspiration prior to the data cutoff date for the analysis.
Time Frame: Median (min, max) follow-up time was 6.3 (2.4, 13.6) months for Phase 1b and 26.7 (3.0, 28.5) months for Phase 2.
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b: Blinatumomab 9/28 μg/Day (Adults) | Phase 1b: Blinatumomab 5/15 µg/m²/Day (Pediatric) | Phase 2: Blinatumomab 9/28 μg/Day (Adults)
Number analyzed (Participants) | 4 | 5 | 8
months | 11.4 [4.2 to 19.7] | 2.3 [1.1 to 6.8] | 13.1 [3.5 to 20.7]

7. Secondary Outcome: Phase 1b and Phase 2: Overall Survival
Description: Overall survival (OS) was calculated from the start date of blinatumomab infusion in the first treatment cycle. All deaths were counted as events on the date of death.
  Participants still alive were censored on the last documented visit date or the date of the last phone contact when the participant was last known to have been alive. For participants who withdrew their informed consent, only information until the date of withdrawal was used in the analysis.
Time Frame: Median (min, max) follow-up time was 6.3 (2.4, 13.6) months for Phase 1b and 26.7 (3.0, 28.5) months for Phase 2.
Population: Phase 1b and Phase 2 participants who received any infusion of blinatumomab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b: Blinatumomab 9/28 μg/Day (Adults) | Phase 1b: Blinatumomab 5/15 µg/m²/Day (Pediatric) | Phase 2: Blinatumomab 9/28 μg/Day (Adults)
Number analyzed (Participants) | 5 | 9 | 21
months | 11.0 [9.3 to 20.7] | 10.6 [0.9 to NA] — could not be estimated due to the low number of events | 14.8 [2.7 to 21.6]

8. Secondary Outcome: Phase 2: Best Overall Response Within 2 Cycles of Treatment
Description: Best response was defined as one of the following:
  CR: ≤ 5% blasts in the bone marrow (BM); No evidence of disease; Full recovery of peripheral blood counts: Platelets > 100,000/µl, and absolute neutrophil count (ANC) > 1,000/µl
  CRh*: ≤ 5% blasts in BM; No evidence of disease; Partial recovery of peripheral blood counts: Platelets > 50,000/µl, and ANC > 500/µl
  CRi: CR with incomplete count recovery without CRh*
  Blast free hypoplastic or aplastic BM: ≤ 5 % blasts in BM; No evidence of disease; Insufficient recovery of peripheral blood counts: platelets ≤ 50,000/µl and/or ANC ≤ 500/µl
  Partial Remission: BM blasts > 5 to < 25% with at least a 50% reduction from baseline
  Hematological Relapse: > 5% blasts in BM or blasts in peripheral blood after documented CR/CRh* during the study
  PD: An increase from baseline of ≥ 25% of BM blasts or an absolute increase of ≥ 5,000 cells/µL in the number of circulating leukemia cells.
Time Frame: Within the first 2 cycles of treatment, 12 weeks
Population: Phase 2 participants who received any infusion of blinatumomab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Blinatumomab 9/28 μg/Day (Adults)
Number analyzed (Participants) | 21
Participants
  CR | 5
  CRh* | 3
  CRi | 0
  Blast-free hypoplastic or aplastic bone marrow | 6
  Partial remission | 0
  Hematological relapse | 0
  PD | 2
  No response (none of the above) | 5

9. Secondary Outcome: Phase 2: Percentage of Participants Who Received an Allogeneic Hematopoietic Stem Cell Transplant (HSCT) During Blinatumomab Induced Remission
Description: Participants who were eligible for allogeneic HSCT were those who achieved remission (complete response or complete response with partial recovery of peripheral blood counts) after 2 cycles of blinatumomab treatment, and no further anti-leukemic medication was given before HSCT.
Time Frame: Median (min, max) follow-up time was 26.7 (3.0, 28.5) months.
Population: Phase 2 participants who received any infusion of blinatumomab.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Blinatumomab 9/28 μg/Day (Adults)
Number analyzed (Participants) | 21
percentage of participants | 81.0

10. Secondary Outcome: Phase 2: 100-Day Mortality After Allogeneic HSCT
Description: The analysis of 100-day mortality after allogeneic HSCT was assessed for all participants who received an allogeneic HSCT while in any CR following treatment with blinatumomab. 100-day mortality after allogeneic HSCT was calculated relative to the date of allogeneic HSCT.
  Participants still alive alive were censored on the last documented visit date or the date of the last phone contact when the patient was last known to have been alive.
  The 100-day mortality rate after allogeneic HSCT was defined as the percentage of participants having died up to 100 days after allogeneic HSCT estimated using the estimated time to death in percent calculated by Kaplan-Meier methods.
Time Frame: 100 days, from the date of allogeneic HSCT; median (min, max) follow-up time was 26.7 (3.0, 28.5)
Population: Phase 2 participants who received an allogeneic HSCT.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Blinatumomab 9/28 μg/Day (Adults)
Number analyzed (Participants) | 17
percentage of participants | 11.8

11. Secondary Outcome: Phase 1b and Phase 2: Number of Participants With TEAEs
Description: TEAEs are defined as those that start between the start of the first infusion of blinatumomab and 30 days after the end of the last infusion during the treatment period.
  The severity of adverse events was assessed by the investigator according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 as follows: Grade 1 - Mild AE; Grade 2 - Moderate AE; Grade 3 - Severe AE; Grade 4 - Life-threatening or disabling AE; Grade 5 - Death.
  The investigator used medical judgment to determine if there was a causal relationship (ie, related, unrelated) between an adverse event and blinatumomab.
Time Frame: From the start of the first infusion to 30 days after the end of the last infusion; median (min, max) treatment duration was 108 (56, 140), 56.0 (5, 84), and 56.0 (11, 115) days in adult phase 1b, adult phase 2 and pediatric phase 1b cohort respectively.
Population: Phase 1b and Phase 2 participants who received any infusion of blinatumomab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Blinatumomab 9/28 μg/Day (Adults) | Phase 1b: Blinatumomab 5/15 µg/m²/Day (Pediatric) | Phase 2: Blinatumomab 9/28 μg/Day (Adults)
Number analyzed (Participants) | 5 | 9 | 21
Participants
  All TEAEs | 5 | 9 | 21
  TEAEs ≥ Grade 3 | 4 | 9 | 21
  TEAEs ≥ Grade 4 | 2 | 7 | 14
  Serious TEAEs (STEAEs) | 0 | 1 | 7
  TEAEs Leading to Blinatumomab Interruption | 1 | 6 | 3
  STEAEs Leading to Blinatumomab Interruption | 0 | 0 | 0
  TEAEs Leading to Blinatumomab Discontinuation | 0 | 1 | 1
  STEAEs Leading to Blinatumomab Discontinuation | 0 | 0 | 1
  Fatal TEAEs | 0 | 1 | 1
  All Treatment-Related (TR) TEAEs | 5 | 8 | 21
  TR TEAEs ≥ Grade 3 | 2 | 8 | 18
  TR TEAEs ≥ Grade 4 | 1 | 5 | 11
  TR STEAEs | 0 | 0 | 4
  TR TEAEs Leading to Blinatumomab Interruption | 1 | 6 | 1
  TR STEAEs Leading to Blinatumomab Interruption | 0 | 0 | 0
  TR TEAEs Leading to Blinatumomab Discontinuation | 0 | 1 | 1
  TR STEAEs Leading to Blinatumomab Discontinuation | 0 | 0 | 1
  TR Fatal TEAEs | 0 | 0 | 0

12. Secondary Outcome: Phase 1b and Phase 2: Serum Blinatumomab Concentration at Steady State
Description: The steady-state concentration (Css) of serum blinatumomab was summarized as the average of the observed concentrations collected after 5 half-lives or after 24 hours from the start of continuous IV infusion.
  Cycle 1, day 2 values represent steady-state concentration after CIV with the initial dose of blinatumomab (9 µg/day for adults and 5 µg/m²/day for pediatric patients). All other time points were measured after the dose step to 28 µg/day (adults) / 15 µg/m²/day (pediatric participants).
Time Frame: After 24 hours from the start of infusion: Cycle 1 (before dose step) day 2; Cycle 1 (after dose step) days 15 and 29; Cycle 2 onwards day 8 (pediatric and adult), days 15 and 29 (adult).
Population: Phase 1b and phase 2 participants who received any infusion of blinatumomab and had at least one pharmacokinetic sample collected, with available data at each time point.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Blinatumomab 9/28 μg/Day (Phase 1b and Phase 2 Adults); Blinatumomab 9/28 μg/Day (Phase 1b Only Adults): Participants received blinatumomab by CIV infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose was 9 μg/day for the first week of cycle 1, escalated to 28 μg/day starting from week 2 and all cycles thereafter.
- Blinatumomab 5/15 µg/m²/Day (Phase 1b and Phase 2 Pediatric); Blinatumomab 5/15 µg/m²/Day (Phase 1b Only Pediatric): Participants received blinatumomab by CIV over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose was 5 µg/m²/day for the first week of cycle 1, escalated to 15 µg/m²/day starting from week 2 and all cycles thereafter.
Arm/Group | Blinatumomab 9/28 μg/Day (Phase 1b and Phase 2 Adults) | Blinatumomab 5/15 µg/m²/Day (Phase 1b and Phase 2 Pediatric) | Blinatumomab 9/28 μg/Day (Phase 1b Only Adults) | Blinatumomab 5/15 µg/m²/Day (Phase 1b Only Pediatric)
Number analyzed (Participants) | 25 | 7 | 5 | 7
pg/mL
  Cycle 1 before dose step: number analyzed (Participants) | 23 | 7 | 4 | 7
  Cycle 1 before dose step | 191 (90.8) | 113 (65.0) | 135 (41.7) | 107 (42.7)
  Cycle 1 after dose step | 948 (488) | 361 (137) | 907 (403) | 361 (137)
  Cycle 2: number analyzed (Participants) | 21 | 6 | 5 | 6
  Cycle 2 | 1150 (575) | 427 (66.0) | 1040 (493) | 427 (66.0)
  Cycle 3+: number analyzed (Participants) | 8 | 1 | 4 | 0
  Cycle 3+ | 1420 (685) | 780 (NA) — could not be calculated for a sample size of 1 | 1280 (396) |

13. Secondary Outcome: Phase 1b and Phase 2: Systemic Clearance of Blinatumomab
Description: Systemic clearance (CL) was calculated as CL = R0/Css, where R0 is the infusion rate (µg/hour or µg/m²/hour).
Time Frame: as for outcome 12
Population: Phase 1b and phase 2 participants who received any infusion of blinatumomab and had at least one pharmacokinetic sample collected.
Measure: Mean (Standard Deviation); unit: liters/hour
Arm/Group | Blinatumomab 9/28 μg/Day (Phase 1b and Phase 2 Adults) | Blinatumomab 5/15 µg/m²/Day (Phase 1b and Phase 2 Pediatric) | Blinatumomab 9/28 μg/Day (Phase 1b Only Adults) | Blinatumomab 5/15 µg/m²/Day (Phase 1b Only Pediatric)
Number analyzed (Participants) | 26 | 9 | 5 | 9
liters/hour | 1.59 (0.812) | 1.88 (0.789) | 1.59 (0.998) | 1.83 (0.801)

14. Secondary Outcome: Phase 1b and Phase 2: Terminal Half-life of Blinatumomab
Time Frame: Cycle 1 day 1 predose, 2, 6 (adults), 10, 24 hours; day 8 (prior to dose step) 0 hour (adults); day 15 any time during infusion; day 29 prior to end of infusion, 1 (adults), 2, 4 (adults), 6 hours after end of infusion
Population: Phase 1b and phase 2 participants who received any infusion of blinatumomab and had at least one pharmacokinetic sample collected with available data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Blinatumomab 9/28 μg/Day (Phase 1b and Phase 2 Adults) | Blinatumomab 5/15 µg/m²/Day (Phase 1b and Phase 2 Pediatric) | Blinatumomab 9/28 μg/Day (Phase 1b Only Adults) | Blinatumomab 5/15 µg/m²/Day (Phase 1b Only Pediatric)
Number analyzed (Participants) | 24 | 5 | 5 | 5
hours | 2.38 (1.36) | 1.92 (1.12) | 2.60 (2.03) | 2.62 (1.67)

15. Secondary Outcome: Phase 1b and Phase 2: Volume of Distribution of Blinatumomab
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Blinatumomab 9/28 μg/Day (Phase 1b and Phase 2 Adults) | Blinatumomab 5/15 µg/m²/Day (Phase 1b and Phase 2 Pediatric) | Blinatumomab 9/28 μg/Day (Phase 1b Only Adults) | Blinatumomab 5/15 µg/m²/Day (Phase 1b Only Pediatric)
Number analyzed (Participants) | 24 | 5 | 5 | 5
liters | 6.02 (6.09) | 5.05 (3.35) | 8.22 (11.7) | 6.38 (3.95)

16. Secondary Outcome: Phase 1b and Phase 2: Number of Participants Who Developed Anti-Blinatumomab Antibodies
Description: Antibodies to blinatumomab were detected using an electrochemiluminescence (ECL)-based assay.
Time Frame: Day 1 before first dose; cycles 1 and 2 day 29, 6 hours after end of infusion; 30 days after last dose.
Population: Phase 1b and Phase 2 participants who received any infusion of blinatumomab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Blinatumomab 9/28 μg/Day (Adults) | Phase 1b: Blinatumomab 5/15 µg/m²/Day (Pediatric) | Phase 2: Blinatumomab 9/28 μg/Day (Adults)
Number analyzed (Participants) | 5 | 9 | 21
Participants | 0 | 0 | 0

17. Secondary Outcome: Phase 1b and Phase 2: Interleukin-2 Concentration
Description: The activation of immune effector cells was monitored by the measurement of peripheral blood cytokine levels including interleukin (IL)-2, IL-6, IL-10, tumor necrosis factor (TNF)-α and interferon gamma (IFN-γ) using multiplex cytometric bead assays. The lower limit of quantification (LLOQ) was 125 pg/mL and the limit of detection (LOD) was 20 pg/mL.
  For calculations of mean cytokine concentrations at every time point across all participants, samples with concentrations below LLOQ were included in the calculation as ½ LLOQ (= 62.5 pg/mL); samples with values below LOD were included as ½ LOD (= 10 pg/mL).
Time Frame: Adults: cycle 1, day 1: 2, 6, 10, 24 hrs after infusion start; day 8: 2, 6, 10 hrs after dose step. Cycles 2-5, day 1: 6 hrs after infusion start. Pediatric: cycle 1, day 1: 6, 10, 24 hrs after infusion start; Cycles 2-5, day 1: 6 hrs after infusion start
Population: Phase 1b and phase 2 participants who received any infusion of blinatumomab and had at least one pharmacodynamic sample collected, with available data at each time point.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Phase 1b and Phase 2: Blinatumomab 9/28 μg/Day (Adults): Participants received blinatumomab by CIV infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose was 9 μg/day for the first week of cycle 1, escalated to 28 μg/day starting from week 2 and all cycles thereafter.
- Phase 1b and Phase 2: Blinatumomab 5/15 µg/m²/Day (Pediatric): Participants received blinatumomab by CIV over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose was 5 µg/m²/day for the first week of cycle 1, escalated to 15 µg/m²/day starting from week 2 and all cycles thereafter.
Arm/Group | Phase 1b and Phase 2: Blinatumomab 9/28 μg/Day (Adults) | Phase 1b and Phase 2: Blinatumomab 5/15 µg/m²/Day (Pediatric)
Number analyzed (Participants) | 26 | 9
pg/mL
  Cycle 1, day 1, 2 hours after start of infusion: number analyzed (Participants) | 26 | 0
  Cycle 1, day 1, 2 hours after start of infusion | 16.1 (17.1) |
  Cycle 1, day 1, 6 hours after start of infusion | 30.2 (72.8) | 10.0 (0.0)
  Cycle 1, day 1, 10 hours after start of infusion | 32.6 (85.0) | 10.0 (0.0)
  Cycle 1, day 1, 24 hours after start of infusion | 17.2 (36.7) | 29.8 (55.9)
  Cycle 1, day 8, 2 hours after start of infusion: number analyzed (Participants) | 25 | 0
  Cycle 1, day 8, 2 hours after start of infusion | 10.0 (0.0) |
  Cycle 1, day 8, 6 hours after start of infusion: number analyzed (Participants) | 25 | 0
  Cycle 1, day 8, 6 hours after start of infusion | 10.0 (0.0) |
  Cycle 1, day 8, 10 hours after start of infusion: number analyzed (Participants) | 25 | 0
  Cycle 1, day 8, 10 hours after start of infusion | 10.0 (0.0) |
  Cycle 2, day 1, 6 hours after start of infusion: number analyzed (Participants) | 20 | 7
  Cycle 2, day 1, 6 hours after start of infusion | 12.6 (11.7) | 10.0 (0.0)
  Cycle 3, day 1, 6 hours after start of infusion: number analyzed (Participants) | 8 | 2
  Cycle 3, day 1, 6 hours after start of infusion | 10.0 (0.0) | 10.0 (0.0)
  Cycle 4, day 1, 6 hours after start of infusion: number analyzed (Participants) | 3 | 1
  Cycle 4, day 1, 6 hours after start of infusion | 10.0 (0.0) | 10.0 (NA) — Could not be calculated for 1 participant
  Cycle 5, day 1, 6 hours after start of infusion: number analyzed (Participants) | 2 | 1
  Cycle 5, day 1, 6 hours after start of infusion | 10.0 (0.0) | 10.0 (NA) — Could not be calculated for 1 participant

18. Secondary Outcome: Phase 1b and Phase 2: Interleukin-6 Concentration
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Phase 1b and Phase 2: Blinatumomab 9/28 μg/Day (Adults) | Phase 1b and Phase 2: Blinatumomab 5/15 µg/m²/Day (Pediatric)
Number analyzed (Participants) | 26 | 9
pg/mL
  Cycle 1, day 1, 2 hours after start of infusion: number analyzed (Participants) | 26 | 0
  Cycle 1, day 1, 2 hours after start of infusion | 29.1 (40.1) |
  Cycle 1, day 1, 6 hours after start of infusion | 173 (198.1) | 275 (371)
  Cycle 1, day 1, 10 hours after start of infusion | 186 (301.5) | 317 (358)
  Cycle 1, day 1, 24 hours after start of infusion | 246 (907.6) | 3714 (10740)
  Cycle 1, day 8, 2 hours after start of infusion: number analyzed (Participants) | 25 | 0
  Cycle 1, day 8, 2 hours after start of infusion | 14.2 (14.5) |
  Cycle 1, day 8, 6 hours after start of infusion: number analyzed (Participants) | 25 | 0
  Cycle 1, day 8, 6 hours after start of infusion | 10.0 (0.0) |
  Cycle 1, day 8, 10 hours after start of infusion: number analyzed (Participants) | 25 | 0
  Cycle 1, day 8, 10 hours after start of infusion | 10.0 (0.0) |
  Cycle 2, day 1, 6 hours after start of infusion: number analyzed (Participants) | 20 | 7
  Cycle 2, day 1, 6 hours after start of infusion | 20.3 (35.6) | 17.5 (19.8)
  Cycle 3, day 1, 6 hours after start of infusion: number analyzed (Participants) | 8 | 2
  Cycle 3, day 1, 6 hours after start of infusion | 16.6 (18.6) | 36.3 (37.1)
  Cycle 4, day 1, 6 hours after start of infusion: number analyzed (Participants) | 3 | 1
  Cycle 4, day 1, 6 hours after start of infusion | 10.0 (0.0) | 62.5 (NA) — Could not be calculated for 1 participant
  Cycle 5, day 1, 6 hours after start of infusion: number analyzed (Participants) | 2 | 1
  Cycle 5, day 1, 6 hours after start of infusion | 10.0 (0.0) | 62.5 (NA) — Could not be calculated for 1 participant

19. Secondary Outcome: Phase 1b and Phase 2: Interleukin-10 Concentration
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Phase 1b and Phase 2: Blinatumomab 9/28 μg/Day (Adults) | Phase 1b: Blinatumomab 5/15 µg/m²/Day (Pediatric)
Number analyzed (Participants) | 26 | 9
pg/mL
  Cycle 1, day 1, 2 hours after start of infusion: number analyzed (Participants) | 26 | 0
  Cycle 1, day 1, 2 hours after start of infusion | 101 (81.1) |
  Cycle 1, day 1, 6 hours after start of infusion | 597 (637) | 153 (94.7)
  Cycle 1, day 1, 10 hours after start of infusion | 423 (373) | 230 (178)
  Cycle 1, day 1, 24 hours after start of infusion | 400 (699) | 641 (1168)
  Cycle 1, day 8, 2 hours after start of infusion: number analyzed (Participants) | 25 | 0
  Cycle 1, day 8, 2 hours after start of infusion | 28.9 (25.7) |
  Cycle 1, day 8, 6 hours after start of infusion: number analyzed (Participants) | 25 | 0
  Cycle 1, day 8, 6 hours after start of infusion | 33.1 (26.6) |
  Cycle 1, day 8, 10 hours after start of infusion: number analyzed (Participants) | 25 | 0
  Cycle 1, day 8, 10 hours after start of infusion | 33.1 (26.6) |
  Cycle 2, day 1, 6 hours after start of infusion: number analyzed (Participants) | 20 | 7
  Cycle 2, day 1, 6 hours after start of infusion | 220 (357) | 142 (173)
  Cycle 3, day 1, 6 hours after start of infusion: number analyzed (Participants) | 8 | 2
  Cycle 3, day 1, 6 hours after start of infusion | 121 (146) | 62.5 (0.0)
  Cycle 4, day 1, 6 hours after start of infusion: number analyzed (Participants) | 3 | 1
  Cycle 4, day 1, 6 hours after start of infusion | 88.2 (93.7) | 62.5 (NA) — Could not be calculated for 1 participant
  Cycle 5, day 1, 6 hours after start of infusion: number analyzed (Participants) | 2 | 1
  Cycle 5, day 1, 6 hours after start of infusion | 36.3 (37.1) | 62.5 (NA) — Could not be calculated for 1 participant

20. Secondary Outcome: Phase 1b and Phase 2: Tumor Necrosis Factor-Alpha (TNFα) Concentration
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Phase 1b and Phase 2: Blinatumomab 9/28 μg/Day (Adults) | Phase 1b and Phase 2: Blinatumomab 5/15 µg/m²/Day (Pediatric)
Number analyzed (Participants) | 26 | 9
pg/mL
  Cycle 1, day 1, 2 hours after start of infusion: number analyzed (Participants) | 26 | 0
  Cycle 1, day 1, 2 hours after start of infusion | 37.3 (61.8) |
  Cycle 1, day 1, 6 hours after start of infusion | 24.1 (23.7) | 15.8 (17.5)
  Cycle 1, day 1, 10 hours after start of infusion | 20.1 (21.1) | 15.8 (17.5)
  Cycle 1, day 1, 24 hours after start of infusion | 10.0 (0.0) | 15.8 (17.5)
  Cycle 1, day 8, 2 hours after start of infusion: number analyzed (Participants) | 25 | 0
  Cycle 1, day 8, 2 hours after start of infusion | 16.6 (32.8) |
  Cycle 1, day 8, 6 hours after start of infusion: number analyzed (Participants) | 25 | 0
  Cycle 1, day 8, 6 hours after start of infusion | 10.0 (0.0) |
  Cycle 1, day 8, 10 hours after start of infusion: number analyzed (Participants) | 25 | 0
  Cycle 1, day 8, 10 hours after start of infusion | 10.0 (0.0) |
  Cycle 2, day 1, 6 hours after start of infusion: number analyzed (Participants) | 20 | 7
  Cycle 2, day 1, 6 hours after start of infusion | 12.6 (11.7) | 17.5 (19.8)
  Cycle 3, day 1, 6 hours after start of infusion: number analyzed (Participants) | 8 | 2
  Cycle 3, day 1, 6 hours after start of infusion | 16.6 (18.6) | 10.0 (0.0)
  Cycle 4, day 1, 6 hours after start of infusion: number analyzed (Participants) | 3 | 1
  Cycle 4, day 1, 6 hours after start of infusion | 10.0 (0.0) | 10.0 (NA) — Could not be calculated for 1 participant
  Cycle 5, day 1, 6 hours after start of infusion: number analyzed (Participants) | 2 | 1
  Cycle 5, day 1, 6 hours after start of infusion | 10.0 (0.0) | 10.0 (NA) — Could not be calculated for 1 participant

21. Secondary Outcome: Phase 1b and Phase 2: Interferon Gamma (IFN-γ) Concentration
Description: as for outcome 17
Time Frame: as for outcome 17
Population: Phase 1b participants who received any infusion of blinatumomab and had at least one pharmacodynamic sample collected, with available data at each time point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Phase 1b and Phase 2: Blinatumomab 9/28 μg/Day (Adults) | Phase 1b and Phase 2: Blinatumomab 5/15 µg/m²/Day (Pediatric)
Number analyzed (Participants) | 26 | 9
pg/mL
  Cycle 1, day 1, 2 hours after start of infusion: number analyzed (Participants) | 26 | 0
  Cycle 1, day 1, 2 hours after start of infusion | 26.2 (24.7) |
  Cycle 1, day 1, 6 hours after start of infusion | 52.3 (56.2) | 41.2 (42.8)
  Cycle 1, day 1, 10 hours after start of infusion | 65.8 (71.6) | 64.5 (107)
  Cycle 1, day 1, 24 hours after start of infusion | 42.1 (51.8) | 129 (176)
  Cycle 1, day 8, 2 hours after start of infusion: number analyzed (Participants) | 25 | 0
  Cycle 1, day 8, 2 hours after start of infusion | 16.3 (17.4) |
  Cycle 1, day 8, 6 hours after start of infusion: number analyzed (Participants) | 25 | 0
  Cycle 1, day 8, 6 hours after start of infusion | 14.2 (14.5) |
  Cycle 1, day 8, 10 hours after start of infusion: number analyzed (Participants) | 25 | 0
  Cycle 1, day 8, 10 hours after start of infusion | 14.2 (14.5) |
  Cycle 2, day 1, 6 hours after start of infusion: number analyzed (Participants) | 20 | 7
  Cycle 2, day 1, 6 hours after start of infusion | 17.9 (19.2) | 40.0 (28.1)
  Cycle 3, day 1, 6 hours after start of infusion: number analyzed (Participants) | 8 | 2
  Cycle 3, day 1, 6 hours after start of infusion | 35.8 (55.0) | 10.0 (0.0)
  Cycle 4, day 1, 6 hours after start of infusion: number analyzed (Participants) | 3 | 1
  Cycle 4, day 1, 6 hours after start of infusion | 10.0 (0.0) | 10.0 (NA) — Could not be calculated for 1 participant
  Cycle 5, day 1, 6 hours after start of infusion: number analyzed (Participants) | 2 | 1
  Cycle 5, day 1, 6 hours after start of infusion | 10.0 (0.0) | 10.0 (NA) — Could not be calculated for 1 participant

22. Primary Outcome: Expansion Cohort: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related TEAEs
Description: as for outcome 11
Time Frame: From the start of the first infusion to 30 days after the end of the last infusion; median (min, max) treatment duration was 55.6 (25, 140) and 28.0 (8, 56) days in the adult and pediatric expansion cohorts, respectively.
Population: Expansion Cohort participants in the who received any infusion of blinatumomab.
Measure: Number; unit: participants
Groups:
- Expansion Cohort: Blinatumomab 9/28 μg/Day (Adults): Participants received blinatumomab by CIV infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose was 9 μg/day for the first week of cycle 1, escalated to 28 μg/day starting from week 2 and all cycles thereafter.
- Expansion Cohort: Blinatumomab 5/15 µg/m²/Day (Pediatric): Participants received blinatumomab by CIV over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose was 5 µg/m²/day for the first week of cycle 1, escalated to 15 µg/m²/day starting from week 2 and all cycles thereafter.
Arm/Group | Expansion Cohort: Blinatumomab 9/28 μg/Day (Adults) | Expansion Cohort: Blinatumomab 5/15 µg/m²/Day (Pediatric)
Number analyzed (Participants) | 14 | 17
participants
  All TEAEs | 14 | 17
  TEAEs ≥ Grade 3 | 11 | 15
  TEAEs ≥ Grade 4 | 7 | 7
  Serious TEAEs (STEAEs) | 2 | 3
  TEAEs Leading to Interruption of Blinatumomab | 2 | 2
  STEAEs Leading to Interruption of Blinatumomab | 0 | 0
  TEAEs Leading to Blinatumomab Discontinuation | 0 | 1
  STEAEs Leading to Blinatumomab Discontinuation | 0 | 0
  Fatal TEAEs | 0 | 2
  All Treatment-Related (TR) TEAEs | 14 | 14
  TR TEAEs ≥ Grade 3 | 9 | 9
  TR TEAEs ≥ Grade 4 | 5 | 5
  TR STEAEs | 0 | 0
  TR TEAEs Leading to Blinatumomab Interruption | 2 | 1
  TR STEAEs Leading to Blinatumomab Interruption | 0 | 0
  TR TEAEs Leading to Blinatumomab Discontinuation | 0 | 1
  TR STEAEs Leading to Blinatumomab Discontinuation | 0 | 0
  TR Fatal TEAEs | 0 | 0

23. Secondary Outcome: Expansion Cohort Adult: Percentage of Participants With a Best Response of Complete Remission or Complete Remission With Only Partial Hematological Recovery Within 2 Cycles of Treatment
Description: as for outcome 2
Time Frame: Within the first 2 cycles of treatment, 12 weeks
Population: Expansion Cohort adult participants who received any infusion of blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Expansion Cohort: Blinatumomab 9/28 μg/Day (Adults)
Number analyzed (Participants) | 14
percentage of participants | 78.6 [49.2 to 95.3]

24. Secondary Outcome: Expansion Cohort Pediatric: Percentage of Participants With M1 Remission Within 2 Cycles of Treatment
Description: as for outcome 4
Time Frame: Within the first 2 cycles of treatment, 12 weeks
Population: Expansion Cohort pediatric participants who received any infusion of blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Expansion Cohort: Blinatumomab 5/15 µg/m²/Day (Pediatric)
Number analyzed (Participants) | 17
percentage of participants | 29.4 [10.3 to 56.0]

ADVERSE EVENTS:
Time Frame: The median treatment duration for blinatumomab was 108 days for Adult Phase 1b Cohort, 56 days for Pediatric Phase 1b Cohort, 56 days for Adult Phase 2 Cohort, 55.6 days for Adult Expansion Cohort and 28 days for Pediatric Expansion Cohort
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Phase 1b: Blinatumomab 9/28 μg/Day (Adults) | Phase 1b: Blinatumomab 5/15 µg/m²/Day (Pediatric) | Phase 2: Blinatumomab 9/28 μg/Day (Adults) | Expansion Cohort: Blinatumomab 9/28 μg/Day (Adults) | Expansion Cohort: Blinatumomab 5/15 µg/m²/Day (Pediatric)
All-Cause Mortality (participants affected / at risk) | 5/5 | 7/9 | 15/21 | 0/14 | 2/17
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/9 | 7/21 | 2/14 | 3/17
Other Adverse Events (participants affected / at risk) | 5/5 | 9/9 | 21/21 | 14/14 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Blinatumomab 9/28 μg/Day (Adults) (N=5) | Phase 1b: Blinatumomab 5/15 µg/m²/Day (Pediatric) (N=9) | Phase 2: Blinatumomab 9/28 μg/Day (Adults) (N=21) | Expansion Cohort: Blinatumomab 9/28 μg/Day (Adults) (N=14) | Expansion Cohort: Blinatumomab 5/15 µg/m²/Day (Pediatric) (N=17)
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Blinatumomab 9/28 μg/Day (Adults) (N=5) | Phase 1b: Blinatumomab 5/15 µg/m²/Day (Pediatric) (N=9) | Phase 2: Blinatumomab 9/28 μg/Day (Adults) (N=21) | Expansion Cohort: Blinatumomab 9/28 μg/Day (Adults) (N=14) | Expansion Cohort: Blinatumomab 5/15 µg/m²/Day (Pediatric) (N=17)
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 7 | 4 | 6
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 7 | 2 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 5 | 10 | 7 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 4 | 3 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 4 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 5 | 5 | 6 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 5 | 3 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Steroid withdrawal syndrome (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 1 | 1 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 8 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 9 | 8 | 2
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 7 | 5 | 2
Vomiting (Gastrointestinal disorders) | 2 | 5 | 3 | 4 | 6
Chest pain (General disorders) | 0 | 0 | 2 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 0 | 0 | 3
Localised oedema (General disorders) | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 1 | 6 | 3 | 0
Oedema (General disorders) | 1 | 1 | 0 | 3 | 0
Pain (General disorders) | 0 | 2 | 0 | 1 | 3
Pyrexia (General disorders) | 1 | 7 | 15 | 4 | 15
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 1 | 4 | 0 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Acute graft versus host disease (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 4 | 5 | 8 | 5 | 6
Hypogammaglobulinaemia (Immune system disorders) | 2 | 2 | 2 | 6 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 3 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 5 | 4 | 2 | 6
Amylase increased (Investigations) | 0 | 2 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 4 | 3 | 0 | 6
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 3 | 1 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 4 | 1 | 1 | 3
Glucose urine present (Investigations) | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 2 | 0 | 0 | 0
Immunoglobulins decreased (Investigations) | 0 | 0 | 3 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 2 | 1 | 1 | 2
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 3 | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 5 | 1 | 3
Oxygen saturation decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 5 | 1 | 5
Prothrombin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Serum ferritin increased (Investigations) | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 1 | 2 | 1 | 2 | 2
White blood cell count decreased (Investigations) | 1 | 1 | 4 | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 3 | 3 | 5
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 3 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 5 | 2 | 0 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 6 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Leukaemic infiltration extramedullary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 4 | 6 | 3 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Intention tremor (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 2 | 1 | 3
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 3 | 3 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 2 | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Asteatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 3 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 4 | 0 | 1 | 2
Hypotension (Vascular disorders) | 1 | 1 | 1 | 0 | 0
Hypoglobulinaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Salivary gland pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Catheter site pain (General disorders) | 0 | 0 | 1 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Engraftment syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Paronychia (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Antithrombin III decreased (Investigations) | 0 | 0 | 0 | 0 | 3
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blast cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood fibrinogen decreased (Investigations) | 0 | 0 | 1 | 0 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Movement disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Wernicke's encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT02412306/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/06/NCT02412306/SAP_001.pdf